CLINICAL TRIAL: NCT03838627
Title: Feasibility and Agreement of Remote Evaluation of Resting Heart Rate and Heart Rate Variability in Survivors of Hodgkin Lymphoma Treated With Chest Radiation (PILOT STUDY-SURVIVOR)
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WHOOPHPP; NCI-2021-05183 (Registry Identifier: NCI)
Record Dates: First submitted 2019-01-23; First posted 2019-02-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Hodgkin Disease
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary Objective The objective is to determine the feasibility and agreement of remote evaluation of resting heart rate and HRV using the commercially available WHOOP® wrist monitor, compared to in-office measurements using AtCor Medical SphygmoCor HRV Software, in a cohort of 40 St. Jude Life Study participants with a history of mantle radiation for management of Hodgkin lymphoma.

Elucidating the mechanisms that contribute to adverse cardiovascular outcomes and reduced quality of life among the growing population of childhood cancer survivors is paramount. Cancer, certain cancer drugs, radiation therapy, cancer-associated lifestyle disturbances, and cancer-independent comorbidities combine to predispose cancer survivors to autonomic dysfunction (AD). Reduced heart rate variability (HRV) has been described in various cancer cohorts. Furthermore, these markers of AD have been implicated in adverse outcomes in oncology patients, including increased mortality, exercise limitation, and fatigue. However, data are largely derived from small studies with methodological limitations, and the contribution of AD to overall morbidity and mortality in cancer survivors is not well understood.

The objective is to determine the feasibility and agreement of remote evaluation of resting heart rate and HRV using the commercially available WHOOP® wrist monitor, compared to in-office measurements using AtCor Medical SphygmoCor HRV Software, in a cohort of 40 St. Jude Life Study participants with a history of mantle radiation for management of Hodgkin lymphoma.

DETAILED DESCRIPTION:
At St. Jude Children's Research Hospital survivors who meet the eligibility criteria will be identified from SJLIFE participants and contacted for potential participation via phone. If the SJLIFE participant expresses interest they will be e-mailed or faxed a copy of the consent form; the consent conference will occur via phone and e-mail or facsimile will be used to document informed consent. Once the consent signature page is received and the participant is enrolled on study, a WHOOP® wrist monitor and directions for wearing the device will be mailed to the participant. Feasibility will be assessed by evaluating how many participants wear and return the device with enough data for analysis. The investigator will consider the project feasible if 30 of 40 participants have 3 hours of usable data after removal of noise. Upon arrival at St. Jude for the St Jude LIFE study, the participant will undergo in-office measurement of HRV while also wearing the WHOOP® device. A standard 10-minute electrocardiogram recording will be performed with the participant in a supine position, with a regular and calm breathing pattern in a quiet room. The standard deviation of normal RR intervals (SDNN, msec) will be derived from SphygmoCor HRV Software. SDNN during this 10-minute time period will be derived from WHOOP® HRV software. Agreement between measures of SDNN derived by the two techniques will be assessed. A mean discrepancy of <20 msec for SDNN measured by the two methods will be considered acceptable agreement.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the SJLIFE study.
* Survivor of childhood Hodgkin lymphoma.
* Exposure to ≥ 20 Gy chest radiation
* Is 18 years of age and older.
* No evidence of cancer recurrence.
* Non-smoker at time of study participation.
* Willingness to avoid caffeine for 3-4 hours and alcohol for 8 hours prior to testing.
* No history of allergic reactions to ECG electrodes.
* Has a smart phone and is willing to download the WHOOP app to their smartphone

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: St. Jude Patients
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The number of patients who wear, return and have sufficient data for analysis of resting heart rate and HRV after removal of noise by WHOOP® HRV software data analysis algorithms. | 48 hours
  Feasibility will be considered adequate if 30 of 40 participants have at least 3 hours of HRV data from the home wearing period.
The degree of agreement between measurements of continuous HRV parameters derived from the two methods will be assessed using linear regression, Pearson's correlation coefficient and Bland Altman analysis. | 10 minute electrocardiogram recording
  A mean discrepancy of <20 msec for SDNN measured by the two methods will be considered acceptable agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten K Ness, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- Kirsten Ness, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Childen's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St.Jude — http://www.stjude.org/protocols

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT03838627/Prot_ICF_000.pdf